CLINICAL TRIAL: NCT00700310
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Study to Evaluate the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Brief Title: Evaluating Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-306; 2007-006169-33 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-11

CONDITIONS: Refractory Partial Seizures
Keywords: Partial onset seizures; E2007; perampanel; refractory partial seizures; adjunctive therapy; seizure frequency; reduction in seizure frequency; safety; concomitant AED(s)
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: perampanel
- 2 (Active Comparator)
  Interventions: Drug: perampanel
- 3 (Active Comparator)
  Interventions: Drug: perampanel
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: perampanel — 2 mg perampanel or placebo in a 1:1:1:1 ratio, 170 subjects/arm, a total of 680 subjects. All subjects will take a maximum of 6 tablets daily and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: E2007
  Arms: 1
Drug: perampanel — 4 mg perampanel or placebo in a 1:1:1:1 ratio, 170 subjects/arm, a total of 680 subjects. All subjects will take a maximum of 6 tablets daily and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: E2007
  Arms: 2
Drug: perampanel — 8 mg perampanel or placebo in a 1:1:1:1 ratio, 170 subjects/arm, a total of 680 subjects. All subjects will take a maximum of 6 tablets daily and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: E2007
  Arms: 3
Drug: Placebo — Placebo in a 1:1:1:1 ratio, 170 subjects/arm, a total of 680 subjects. All subjects will take a maximum of 6 tablets daily.
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of perampanel when given as an adjunctive therapy in subjects with refractory partial seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent signed by the subject or legal guardian prior to entering the study or undergoing any study procedures (If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained.).
2. Be considered reliable and willing to be available for the study period and able to record seizures and report AEs them self or have a caregiver who can record seizures and report AEs for them;
3. Male or female and greater than or equal to 12 years of age (within the course of the study), or greater than or equal to 18 years of age (depending on location) at the time of signing the informed consent.
4. Females should be either of non-childbearing potential (defined as having undergone surgical sterilization, or postmenopausal [age 50 and amenorrheic for 12 months]) or of childbearing potential. Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin (ß-hCG) at Visit 1 and a negative urine pregnancy test prior to randomization at Visit 2. Female subjects of childbearing potential must agree to be abstinent or to use at least 1 medically acceptable methods of contraception (eg, a double-barrier method [eg, condom + spermicide, condom + diaphragm with spermicide], IUD, or have a vasectomised partner) starting at Visit 1 and throughout the entire study period and for 2 months after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously) starting at Visit 1 and continuing throughout the entire study period and for 2 months after the last dose of study drug. (It is not required for male subjects to use contraceptive measures based on preclinical toxicology data.);
5. Have a diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization-related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history);
6. Have had a computed tomography (CT) or magnetic resonance imaging (MRI) within the last 10 years that ruled out a progressive cause of epilepsy;
7. Have uncontrolled partial seizures despite having been treated with at least 2 different anti-epileptic drugs (AEDs) within approximately the last 2 years;
8. During the 6-week Pre-randomization Phase subjects must have had >/= 5 partial seizures per 6-week (with >/=2 partial seizures per each of 3-week period) and with no 25-day seizure-free period in the 6-week period, as documented via a valid seizure diary. Only simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with secondary generalization are counted toward this inclusion;
9. Are currently being treated with stable doses of 1, 2 or a maximum of 3 approved AEDs. Only 1 inducer AED (defined as; carbamazepine, phenytoin, phenobarbital, or primidone only) out of the maximum of 3 AEDs is allowed;
10. Are on a stable dose of the same concomitant AED(s) for 1 month (or no less than 21 days) prior to Visit 1; in the case where a new AED regime has been initiated for a subject, the dose must be stable for 2 months (or no less than 49 days) prior to Visit 1;
11. If on a stable dose (other than intermittent rescue use) of benzodiazepines for epilepsy (or for anxiety or sleep disorders) the prescribed dose must be stable for 1 month (or no less than 21 days) prior to Visit 1. (Note: the use of intermittent rescue benzodiazepines is defined in the exclusion criterion #22 below.) When used in these cases (epilepsy, anxiety or sleep disorders), benzodiazepines will be counted as 1 AED; therefore, only 1 or a maximum of 2 additional approved AEDs will be allowed;
12. A vagal nerve stimulator (VNS) is allowed but it must have been implanted >/= 5 months prior to Visit 1. Stimulator parameters can not be changed for 1 month (or no less than 21 days) prior to Visit 1 or thereafter during the study.

Exclusion Criteria:

1. Participated in a study involving administration of an investigational compound or device within 1 month (or no less than 21 days) prior to Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer;
2. Pregnant and/or lactating;
3. Participated in previous perampanel studies;
4. Presence of nonmotor simple partial seizures only;
5. Presence of primary generalized epilepsies or seizures, such as absences and or myoclonic epilepsies;
6. Presence or previous history of Lennox-Gastaut syndrome;
7. A history of status epilepticus within approximately 12 months prior to Visit 1;
8. Seizure clusters where individual seizures cannot be counted;
9. A history of psychogenic seizures;
10. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the Investigator(s) could affect the subject's safety or the study conduct;
11. Scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1; however those who have previously documented "failed" epilepsy surgery will be allowed;
12. Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than 3 times the upper limit of normal (ULN);
13. Evidence of significant active hematological disease; white blood cell (WBC) count <= 2500/µL (2.50 1E+09/L) or an absolute neutrophil count <= 1000/µL (1.00 1E+09/L);
14. A clinically significant ECG abnormality, including prolonged QTc defined as >450 msec;
15. Suffering from psychotic disorder(s) and/or unstable recurrent affective disorder(s) evident by use of antipsychotics or have had a suicide attempt(s) within the last 2 years.
16. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors;
17. History of drug or alcohol dependency or abuse within approximately the last 2 years;
18. Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions;
19. If felbamate is used as a concomitant AED, subjects must be on felbamate for at least 2 years, with a stable dose for 2 months (or no less than 49 days) prior to Visit 1. They must not have a history of white blood cell (WBC) count below 2500/µL (2.50 1E+09/L), platelets below 100,000, liver function tests (LFTs) above 3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If patients received felbamate in the past, it must have been discontinued 2 months (or no less than 49 days) prior to Visit 1;
20. Concomitant use of vigabatrin. Subjects who took vigabatrin in the past must be off vigabatrin for approximately 5 months prior to Visit 1 and must have documentation showing no evidence of a vigabatrin associated clinically significant abnormality in a visual perimetry test;
21. Concomitant use of barbiturates (except for seizure control indication) within 1 month (or no less than 21 days) prior to Visit 1;
22. Use of intermittent rescue benzodiazepines (ie, 1-2 doses over a 24-hr period considered one-time rescue) 2 or more times in a 1-month period prior to Visit 1; or
23. Any condition(s) that will make the subject, in the opinion of the Investigator, unsuitable for the study.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (108):
- Australia (11):
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Woodville South, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - Parkville, Victoria
  - Clayton
  - Fitzroy
  - Parkville
  - West Heidelberg
  - Woodville
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Germany (8):
  - Düsseldorf
  - Kehl-Kork
  - Konigstein-Falkenstein
  - Mainz
  - Marburg
  - München
  - Ulm
  - Westerstede
- Hong Kong (6):
  - Queen Mary Hospital, Hong Kong
  - Hong Kong
  - Queen Elizabeth Hospital, Kowloon
  - United Christian Hospital, Kowloon
  - Kowloon
  - Prince of Wales Hospital, Shatin
- Hungary (2):
  - Budapest
  - Kecskemét
- India (6):
  - Hyderabad, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Jaipur, Rajasthan
  - New Delhi
- Italy (5):
  - Milan
  - Napoli
  - Padua
  - Siena
  - Torino
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Malaysia (2):
  - Kuala Lumpur, Kuala Lumpur
  - Kuala Terengganu, Terengganu
- Philippines (2):
  - Ermita
  - Makati City
- Poland (7):
  - Bialystok
  - Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Katowice
  - Lodz
  - Lublin
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Romania (7):
  - Brasov
  - Sapiens Medical Center, Bucharest
  - Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Pediatric Neurology Clinic of Emergency Children Hospital, Cluj-Napoca
  - Cluj-Napoca
- Russia (8):
  - Moscow State University of Medicine and Dentistry, Moscow
  - Moscow
  - Moscow Research Institute of Psychiatry, Moscow
  - Moscow Research Institute of Pediatrics and Pediatric Surgery, Moscow
  - Samara
  - Tyumen
  - Yaroslavl
  - Yekaterinburg
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad
- South Korea (3):
  - Busan
  - Daegu
  - Seoul
- Spain (8):
  - Granada, Andalusia
  - Badalona, Catalonia
  - Barcelona, Catalonia
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Valencia, Valencia
  - Barcelona
  - Valencia
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taoyuan District
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Muang District
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Uzhhorod

REFERENCES:
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] French JA, Gil-Nagel A, Malerba S, Kramer L, Kumar D, Bagiella E. Time to prerandomization monthly seizure count in perampanel trials: A novel epilepsy endpoint. Neurology. 2015 May 19;84(20):2014-20. doi: 10.1212/WNL.0000000000001585. Epub 2015 Apr 15. PMID 25878175
- [Derived] Rosenfeld W, Conry J, Lagae L, Rozentals G, Yang H, Fain R, Williams B, Kumar D, Zhu J, Laurenza A. Efficacy and safety of perampanel in adolescent patients with drug-resistant partial seizures in three double-blind, placebo-controlled, phase III randomized clinical studies and a combined extension study. Eur J Paediatr Neurol. 2015 Jul;19(4):435-45. doi: 10.1016/j.ejpn.2015.02.008. Epub 2015 Mar 5. PMID 25823975
- [Derived] Steinhoff BJ, Ben-Menachem E, Ryvlin P, Shorvon S, Kramer L, Satlin A, Squillacote D, Yang H, Zhu J, Laurenza A. Efficacy and safety of adjunctive perampanel for the treatment of refractory partial seizures: a pooled analysis of three phase III studies. Epilepsia. 2013 Aug;54(8):1481-9. doi: 10.1111/epi.12212. Epub 2013 May 10. PMID 23663001
- [Derived] Krauss GL, Serratosa JM, Villanueva V, Endziniene M, Hong Z, French J, Yang H, Squillacote D, Edwards HB, Zhu J, Laurenza A. Randomized phase III study 306: adjunctive perampanel for refractory partial-onset seizures. Neurology. 2012 May 1;78(18):1408-15. doi: 10.1212/WNL.0b013e318254473a. Epub 2012 Apr 18. PMID 22517103

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo over 19-weeks (during 6-week Titration phase and 13-week Maintenance phase)
- Perampanel 2mg: Perampanel 2mg daily over 19-weeks (during 6-week Titration phase and 13-week Maintenance phase)
- Perampanel 4mg: Perampanel 4mg maximum daily dose (Titration from 2mg to 4mg daily over 6-weeks; Maintenance at 4 mg daily over 13-weeks)
- Perampanel 8 mg: Perampanel 8mg maximum daily dose (Titration from 2mg to 8mg daily over 6-weeks; Maintenance at 8 mg daily over 13-weeks)
Period: Overall Study
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg
Started | 187 | 180 | 174 | 171
Completed | 166 | 154 | 158 | 145
Not Completed | 21 | 26 | 16 | 26
Not completed — Adverse Event | 6 | 10 | 5 | 11
Not completed — Lost to Follow-up | 4 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 9 | 8 | 8
Not completed — Lack of Efficacy | 0 | 3 | 0 | 1
Not completed — Administrative/Other | 1 | 3 | 1 | 3
Not completed — Randomized, Not Treated | 2 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg | Total
Number analyzed (Participants) | 185 | 180 | 172 | 169 | 706
Age, Customized [Number; unit: Participants]
  <18 Years | 14 | 21 | 13 | 12 | 60
  18-64 Years | 169 | 156 | 158 | 153 | 636
  >64 Years | 2 | 3 | 1 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — The number of participants started is not consistant with the number of Baseline Participants due to 6 participants who were randomized in the study, but not treated with study drug.
  Participants
    Female | 90 | 95 | 84 | 92 | 361
    Male | 95 | 85 | 88 | 77 | 345
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 119 | 119 | 105 | 116 | 459
    Asian | 34 | 35 | 37 | 28 | 134
    Chinese | 31 | 25 | 29 | 25 | 110
    Other | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full Intent-to-Treat (ITT) Analysis Set - group of subjects who were randomized to study drug, received study drug, and had any seizure frequency data during the Double-blind Phase.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg
Number analyzed (Participants) | 184 | 180 | 172 | 169
Percent Change | -10.69 [-100.0 to 420.6] | -13.63 [-100.0 to 346.3] | -23.33 [-100.0 to 416.0] | -30.80 [-100.0 to 390.6]

2. Secondary Outcome: Responder Rate
Description: The responder rate for the Full ITT Analysis Set from the maintenance LOCF (Last Observation Carried Forward). A responder was a subject who had a 50 percent or greater reduction in seizure frequency per 28 days from the Pre-randomization phase.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg
Number analyzed (Participants) | 184 | 180 | 172 | 169
Percentage of Participants
  Responders (Yes) | 17.9 | 20.6 | 28.5 | 34.9
  Non-Responders (No) | 82.1 | 79.4 | 71.5 | 65.1

3. Secondary Outcome: Percent Change in the 28-day Complex Partial Plus Secondarily Generalized Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Percent Change in the Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg
Number analyzed (Participants) | 169 | 167 | 157 | 154
Percent Change | -17.63 [-100.0 to 602.9] | -20.50 [-100.0 to 13744.2] | -31.18 [-100.0 to 416.0] | -38.69 [-100.0 to 583.3]

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent form to 30 days after the last dose of the study drug.
Description: Adverse events were assessed at clinical visits based on the subject's diary, vitals, weight, physical examination, neurological exam, and laboratory evaluations; and by telephone interviews/contact.
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 8 mg
Serious Adverse Events (participants affected / at risk) | 9/185 | 6/180 | 6/172 | 6/169
Other Adverse Events (participants affected / at risk) | 48/185 | 61/180 | 66/172 | 79/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=185) | Perampanel 2mg (N=180) | Perampanel 4mg (N=172) | Perampanel 8 mg (N=169)
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 3 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0
Simple partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=185) | Perampanel 2mg (N=180) | Perampanel 4mg (N=172) | Perampanel 8 mg (N=169)
Fatigue (General disorders) | 5 | 8 | 13 | 9
Gait disturbance (General disorders) | 2 | 1 | 2 | 9
Nasopharyngitis (Infections and infestations) | 3 | 7 | 9 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 11 | 6 | 3
Dizziness (Nervous system disorders) | 18 | 18 | 28 | 45
Headache (Nervous system disorders) | 16 | 16 | 19 | 18
Somnolence (Nervous system disorders) | 12 | 22 | 15 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No